CLINICAL TRIAL: NCT06410456
Title: The Effect of Schroth Exercises on Cerebral Cortical Thickness and Motor and Proprioceptive Fibres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Ahmet Payas, Assistant professor, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 932
Record Dates: First submitted 2024-03-17; First posted 2024-05-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth exercises groups (Experimental): Adolescents with idiopathic scoliosis received Schroth exercises four days a week for six months.
  Interventions: Other: Schroth exercises
- Traditional exercises groups (Experimental): Adolescent idiopathic scoliosis patients underwent stretching exercises (especially for the muscles on the concave side of the curve), posture training, strengthening and spinal flexibility exercises as conventional exercises four days a week for six months.
  Interventions: Other: Traditional exercises

INTERVENTIONS:
Other: Schroth exercises — Traditional exercise
  Arms: Schroth exercises groups
Other: Traditional exercises — Adolescents with idiopathic scoliosis performed conventional exercises four days a week for six months.
  Arms: Traditional exercises groups

SUMMARY:
Adolescent idiopathic scoliosis (AIS): It is a type of structural scoliosis of unknown aetiology and most commonly seen in girls aged 10-18 years. In addition to spinal deformity, postural asymmetry, proprioceptive sensory, vestibular and vestibulospinal system dysfunctions may be observed in AIS. The Schroth method is a scoliosis-specific exercise approach that uses postural, scoliosis-specific sensorimotor and breathing exercises and is widely used in scoliosis rehabilitation. The treatment programme consists of correction of scoliotic posture with the help of exteroceptive and proprioceptive stimulation and mirrors, isometrics and other exercises to lengthen or strengthen asymmetric muscles, and maintaining a specific breathing pattern. Several studies have shown that the Schroth method improves Cobb angles, slows curve progression, reduces the need for surgery, increases back muscle strength and improves respiratory function. However, although the Schroth method is widely used in AIS rehabilitation, no study has investigated the effects of Schroth exercises on cerebral cortical thickness, proprioceptive sensation and corticospinal pathways.

The aim of this study was to compare the effects of Schroth and traditional exercises on cortical thickness, proprioceptive sensation and corticospinal tracts in individuals with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Being a female individual between the ages of 10-18
* Being diagnosed with AIS
* Cobb angle should be maximum 25º
* All participants do not have any disease that affects the nervous system.
* All participants must use their right hand as the dominant hand
* All participants do not have any chronic disease requiring the use of any neurological or psychiatric medication.
* Permission to participate in the study is given by the parents of all participants.

Exclusion Criteria:

* MRI of individuals who do not have any mental problems, neurological, psychiatric, muscular, rheumatic or orthopedic diseases will be included in the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Tractography | Six months
  Number of fibers of tractus corticospinalis, lemniscus medialis tracts
VolBrain | Six months
  Brain cortical thickness measurement
Cobb angle | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Payas, Ph.D, Study Director — Amasya University
Locations (1):
- Ahmet Payas, Kayseri, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Result] Kocaman H, Bek N, Kaya MH, Buyukturan B, Yetis M, Buyukturan O. The effectiveness of two different exercise approaches in adolescent idiopathic scoliosis: A single-blind, randomized-controlled trial. PLoS One. 2021 Apr 15;16(4):e0249492. doi: 10.1371/journal.pone.0249492. eCollection 2021. PMID 33857180
- [Result] Li P, Legault J, Litcofsky KA. Neuroplasticity as a function of second language learning: anatomical changes in the human brain. Cortex. 2014 Sep;58:301-24. doi: 10.1016/j.cortex.2014.05.001. Epub 2014 May 17. PMID 24996640
- [Result] Sagi Y, Tavor I, Hofstetter S, Tzur-Moryosef S, Blumenfeld-Katzir T, Assaf Y. Learning in the fast lane: new insights into neuroplasticity. Neuron. 2012 Mar 22;73(6):1195-203. doi: 10.1016/j.neuron.2012.01.025. Epub 2012 Mar 21. PMID 22445346
- [Derived] Payas A, Kocaman H, Yildirim H, Arik M, Batin S. Associations Between Different Exercise Approaches and Brain Structure in Adolescent Idiopathic Scoliosis: An Exploratory Neuroimaging Study. Global Spine J. 2025 Dec 22:21925682251411247. doi: 10.1177/21925682251411247. Online ahead of print. PMID 41424174